CLINICAL TRIAL: NCT04819412
Title: A Seamless, Sequential Phase III, Randomized, Multi Center Single Blind Study to Evaluate Immunogenicity, Safety, Reactogenicity of Liquid ROTAVAC 5C Vaccine as a 3-dose Series When Compared With ROTAVAC® in Infants
Brief Title: To Determine the Safety and Efficacy of Liquid ROTAVAC 5C Vaccine Against Childhood Diarrhea Caused by Rotavirus
Acronym: ROTAVAC5C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Collaborators: Georgia Institute for Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BBIL/ROTA5C/III/2014
Record Dates: First submitted 2020-07-11; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Rotavirus Gastroenteritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ROTAVAC 5C -F1 (Experimental): ROTAVAC 5C formulation BBIL-R2014-1
  Interventions: Biological: ROTAVAC 5C -F1
- ROTAVAC 5C -F2 (Experimental): ROTAVAC5C formulation BBIL-R2014-2
  Interventions: Biological: ROTAVAC 5C -F2
- ROTAVAC® (Active Comparator): ROTAVAC® with 5 minutes prior administration of 2.5 ml of buffer
  Interventions: Biological: ROTAVAC®

INTERVENTIONS:
Biological: ROTAVAC® — ROTAVAC® with 5 minutes prior administration of 2.5 ml of buffer
  Arms: ROTAVAC®
Biological: ROTAVAC 5C -F1 — ROTAVAC 5C formulation BBIL-R2014-1
  Arms: ROTAVAC 5C -F1
Biological: ROTAVAC 5C -F2 — ROTAVAC 5C formulation BBIL-R2014-2
  Arms: ROTAVAC 5C -F2

SUMMARY:
Study Rationale A single Rotavirus vaccine container with the vaccine virus and antacid buffer would be ideal for logistical, administrative and distribution ease, especially in routine immunization program.

* The advantages of the liquid vaccines are: Liquid vaccines take lesser time to administer compared to the current practice of giving antacid buffer prior to vaccine which takes 40% more time to administer.
* Easier to transport as it is stable at 2-80C compared to the frozen formulation that needs to be stored at -200C and transported in dry ice.
* Chances of human error during administration are lesser than the sequential administration of antacid and vaccine.

DETAILED DESCRIPTION:
Study Design and plan The study is designed as an adaptive, seamless sequential multicenter, single-blinded, randomized clinical trial with two phases: exploratory phase and confirmatory phase.

Exploratory phase:

1. Infants of 6-8 weeks of age will randomly be assigned to receive 3 doses of two different formulations of ROTAVAC 5C (BBIL-R2014-1 &BBILR2014-2) or ROTAVAC®. In this phase, immunogenicity and safety of the two new formulations will be compared with each other and with ROTAVAC® in the three treatment arms when administered at 4 weeks interval (+1week window). The first dose will be administered at 6-8 weeks of age. Each of the rotavirus vaccine formulations contains NLT 105fluorescent focus units (FFU)/Dose. After completion of the exploratory phase, analyses will be undertaken for selection of the most suitable formulation to undergo confirmatory phase of the study.

Confirmatory Phase:

1. Infants of 6-8 weeks of age will randomly be assigned to receive 3 doses of the selected formulation of ROTAVAC 5C (3 production lots) and ROTAVAC® to evaluate lot consistency. Additionally, non-interference with immune response to antigens contained in childhood vaccines will be evaluated.
2. Active surveillance will be conducted for all participants for seven days after each dose of vaccine to ascertain information on solicited adverse events.("Reactogenicity")
3. Surveillance for unsolicited AEs for all participants will be conducted from the time between first dose and 4-6 weeks after the 3rd dose.

Surveillance for SAEs for all participants will be conducted from the time between first dose and 4-6 weeks after the 3rd dose

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as established by medical history and clinical examination before entering the study.
2. Age: 6-8 weeks
3. Weight ≥2.5 kgs at birth.
4. Infants received EPI vaccines (OPV, BCG and Hep B) at birth.
5. Parental ability and willingness to provide informed consent.
6. Parent who intends to remain in the area with the participant during the study period.

   -

Exclusion Criteria:

1. Presence of diarrhoea or vomiting in the previous 72 hours or on the day of enrolment (temporary exclusion).
2. Presence of fever on the day of enrolment (temporary exclusion).
3. Concurrent participation in another clinical trial.
4. Presence of significant malnutrition or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, immuno-logical, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination which would compromise the child's health or is likely to result in non-conformance to the protocol.
5. History of congenital abdominal disorders, intussusception, abdominal surgery
6. Known or suspected impairment of immunological function based on medical history and physical examination.
7. Household contact with an immunosuppressed individual or pregnant woman.
8. Prior receipt of rotavirus vaccine.
9. A known sensitivity or allergy to any components of the study vaccines.
10. Major congenital or genetic defect.
11. History of persistent diarrhoea (defined as diarrhoea more than 14 days).
12. Participant's parents not able, available or willing to accept active follow-up by the study staff.
13. Has received any immunoglobulin therapy and/or blood products since birth.
14. History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
15. History of any neurologic disorders or seizures.
16. Any medical condition in the parents/infants that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parent's/legally acceptable representative's ability to give informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1975 (Actual)
Dates: Start 2015-03-20; Primary Completion 2015-10-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity in terms of GMT and four-fold seroconversion | from Baseline 84 days.
  Immunogenicity

SECONDARY OUTCOMES:
Occurrence of adverse events and Serious Adverse events | from base line to 84 days
  safety
Evaluation of shedding of rotavirus. | Stool specimen: Day 3 and 7 after each vaccine dose
  Viral shedding